CLINICAL TRIAL: NCT06210230
Title: Double-blind and Placebo-controlled Study on Intervention Effect of Medium and Long Chain Fatty Acid Triglyceride on Glycolipid Homeostasis in Patients With Metabolic Syndrome and Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Yu Zhang, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT_MLCT_MetS
Record Dates: First submitted 2024-01-06; First posted 2024-01-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-05

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; MLCT
MeSH Terms: conditions — Metabolic Syndrome | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Dietary Supplement: Olive oil
- Intervention group (Experimental)
  Interventions: Dietary Supplement: MLCT supplementation

INTERVENTIONS:
Dietary Supplement: MLCT supplementation — MLCT 25g/d for 6 months
  Arms: Intervention group
Dietary Supplement: Olive oil — Matching placebo (olive oil) 25g/d for 6 months
  Arms: Control group

SUMMARY:
Double-blind and placebo-controlled study on intervention effect of medium and long chain fatty acid triglyceride on glycolipid homeostasis in patients with metabolic syndrome and mechanisms

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed metabolic syndrome according to IDF diagnostic criteria;
* Rarely eating out of home;
* Aged between 40 and 70 years.

Exclusion Criteria:

* Breastfeeding or pregnancy;
* History of heart disease, coronary heart disease, stroke, cerebral infarction, viral liver disease (hepatitis A, hepatitis B, etc.), chronic kidney disease (GFR<60 ml/min) or cancer;
* Diabetic ketoacidosis or hyperketosis;
* Drug use has changed in the past six months;
* Taking insulin;
* Used MLCT edible oil in the past six months;
* Have participated in other clinical trials in the last three months.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose from baseline | 6 months
  The investigators will measure HbA1c and fasting plasma glucose levels in blood samples before and after treatment.
Change in blood lipids from baseline | 6 months
  The investigators will measure Triglycerides (TG), total cholesterol (TC), LDL-C, and HDL-C levels in blood samples before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Lanxi Traditional Chinese Medicine Hospital, Jinhua, Zhejiang, China